CLINICAL TRIAL: NCT03088215
Title: Treating Fibromyalgia Pain With Shock-Waves: a Randomized Study
Brief Title: Shock-Waves to Treat Fibromyalgia Pain
Acronym: SWPW-FPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr Yves JACOT, MD (Other)
Collaborators: Projet Suisse d'Assistance Medicale (Other)
Responsible Party: Sponsor-Investigator, Dr Yves JACOT, MD, Director, Projet Suisse d'Assistance Medicale
Organization: Projet Suisse d'Assistance Medicale (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWPW-FPS - v1.0 - 07/03/2017
Record Dates: First submitted 2017-03-10; First posted 2017-03-23 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Fibromyalgia; Myofascial Pain Syndrome; MSK: Chronic Pain Syndromes (E.G. Fibromyalgia); Central Sensitization
Keywords: Trigger Point Pain, Myofascial; shock-waves; extracorporeal shock-wave treatment (ESWT); pain; trigger point; referred pain
MeSH Terms: conditions — Fibromyalgia; Myofascial Pain Syndromes; Pain; Pain, Referred

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A / Shock-waves (Experimental): Will receive shock-waves
  Interventions: Device: shock-waves
- B / Nothing (No Intervention): Will not receive shock-waves

INTERVENTIONS:
Device: shock-waves — Application of shock-waves (radial and focused)
  Arms: A / Shock-waves

SUMMARY:
Fibromyalgia pain syndrome is a common debilitating condition which associates mainly generalised pain, emotional distress and cognitive symptoms. The etiology is unknown, and no specific treatment exists so far.

Lately, shock-waves have been used successfully to treat painful skeletal muscle, tendons and fascia, the investigators therefore hypothesize that shock-waves could be useful in alleviating Fibromyalgia pain.

Two similar groups of participants bearing the condition will be prospectively compared.

The first group will benefit from the application of shock-waves weekly for 12 weeks, the second will not.

The investigators intend to study if there is any difference in pain and quality of life between the two groups at the end of the three months.

DETAILED DESCRIPTION:
Fibromyalgia Pain Syndrome (FPS) is a common debilitating condition which associates mainly generalised pain, emotional distress and cognitive symptoms. The etiology is unknown, and no specific treatment exists so far.

It bears some similarities with another, more localised clinical condition : the Myofascial Pain Syndrome (MPS), which results in pain caused by, amongst others, muscular trigger points.

Lately, FPS and MPS have both been classified as belonging to a new, larger entity : Central Sensitivity Syndromes (CSS), in which a strong and chronic peripheral sensitive stimulus (like musculoskeletal pain) is believed to induce, after some time, an enhanced response of the central nervous system (CNS) towards that same stimulus, with the result that the stimulus will be felt more powerfully (central sensitization, CS). This is secondary to neuroplastic changes in the CNS, which are reversible to some extent.

Since shock-waves are effective to treat pain in MPS (by eliminating trigger points and thus restoring muscle and tissue function), and since MPS and FPS could be linked by a common pathophysiologic mechanism (CSS), the investigators hypothesize that shock waves could be beneficial in treating pain in FPS.

Two groups of 20 participants will be prospectively compared over a three month's period.

One group will receive shock-waves on painful muscular areas weekly for 12 weeks, the other group will not receive any shock-waves.

The investigators intend to study if there is any difference in pain and quality of life after the end of the three months.

ELIGIBILITY:
Inclusion Criteria:

* American College of Rheumatology 2011 diagnostic criteria for Fibromyalgia met
* Aged between 18 and 65 years
* Informed Consent Form signed

Exclusion Criteria:

* Known skeletal pathologies such as osteoarthritis of major joints and / or vertebrae, inflammatory states involving bones, joints, tendons or muscles, or previous heavy trauma directly causing the pain
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, carcinoma, cardiovascular disease, pulmonary insufficiency, etc.),
* Coagulopathies, anticoagulant or corticosteroid based medication, thrombosis.
* Psychological distress, psychosis, dementia
* Known or suspected non-compliance, drug or alcohol abuse,
* Pregnancy
* Enrolment of the investigator, his/her family members, employees and other dependent or vulnerable persons

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-10-20 (Estimated); Primary Completion 2018-11-20 (Estimated); Study Completion 2018-11-20 (Estimated)

PRIMARY OUTCOMES:
Pain VAS | 12 weeks
  Horizontal visual analog scale for pain (pain intensity)

SECONDARY OUTCOMES:
Apparent change in successive Pain Body Maps over time | 12 weeks
  Participants will be distributed successive body map models where they are asked to draw the precise location and extension of the areas where they experience pain.
  The maps completed at every given time will then be compiled for each group (by computer).
  The final compiled pictures will be visually compared between each group. So far, it is not planned to do measurements (such as surface, etc...), the maps will serve mainly illustrate differences in pain extension between the two groups.
Interference scale of the Body Pain Index (BPI) | 12 weeks
  Questionnaire reflecting interference of pain in quality of life
Patient Global Impression of Change scale (PGIC) | 12 weeks
  Questionnaire reflecting effects of intervention (or non-intervention)from the participant's point of view

OTHER OUTCOMES:
American College of Rheumatology (ACR) diagnostic criteria 2011 for Fibromyalgia | 12 weeks
  Serves to assess if participants in intervention arm still meet the diagnostic criteria for Fibromyalgia at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Dr Yves JACOT, MD, Study Director

IPD SHARING:
Plan to Share IPD: Undecided